CLINICAL TRIAL: NCT06289296
Title: Metabolic Effects of Dietary Medium-Chain Fatty Acids.
Brief Title: Medium Chain Fatty Acids and Ketones
Acronym: MCFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Kiens, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MCT
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Diet, Healthy; Health
Keywords: medium-chain fatty acids; ketones; Obesity
MeSH Terms: conditions — Ketosis; Obesity

STUDY DESIGN:
Intervention Model Description: A parallel crossover design, in which a group of lean and a group of obese participants are allocated to complete two seven-day intervention periods with twice daily consumption of either medium-chain fatty acids or long-chain fatty acids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fatty acid intake in lean males (Experimental): Lean males will be studied before and after 7 days daily intake of either Medium-chain fatty acids or Long-chain fatty acids. . After a wash-out period the intervention is repeated in opposite sequence.
  Interventions: Other: Fatty acid intake in lean and obese males
- Fatty acid intake in obese males (Experimental): In obese male participants will be studied before and after 7 days daily intake of either medium-chain fatty acids (MCT) or long-chain fatty acids (LCT). After a wash-out period the intervention is repeated in opposite sequence.
  Interventions: Other: Fatty acid intake in lean and obese males

INTERVENTIONS:
Other: Fatty acid intake in lean and obese males — Acute and chronic intake of MCT and LCT

SUMMARY:
16 participants were randomized to complete two seven-day intervention periods with twice-daily consumption of Medium-chain fatty acids (MCT) or long-chain fatty acids (LCT) oil. Before and after each intervention, participants completed a five-hour experimental day evaluating the response to a first intake of the MCT or LCT oils (pre MCT or LCT), which was repeated after the intervention period of daily intake (post MCT or LCT) (Fig. The intervention periods were separated by a 2-4-week washout period.

DETAILED DESCRIPTION:
Prior to the experimental days, the participants abstained from alcohol and vigorous physical activity and consumed a controlled, eucaloric diet comprising 30 energy % (E%) fat, 52 E% carbohydrate, and 18E% protein to ensure similar conditions before each experimental day.

On the experimental days, participants arrived by passive transport in the overnight fasted state (12 h) at 8 a.m at the institute. At arrival, participants were weighed, and body composition was determined using dual-energy x-ray absorptiometry (DXA). Then a catheter was inserted into an antecubital vein. Following 30 min of supine rest, whole-body oxygen uptake and substrate oxidation were determined, whereafter a basal venous blood sample was obtained. Subsequently, participants ingested a test drink containing 35g of MCT or LCT oil diluted in 100g of a low-fat, low-carbohydrate cocoa milk within five min. 100 ml water was provided together with the test drink. Participants were blinded to the type of oil intake on the experimental days. The participants were then followed for five hours. Venous blood samples and indirect calorimetry measurements were performed frequently during the five hours. Participants rested in a bed throughout the test day.

Following the first test day, a seven-day intervention period (chronic intake) with twice-daily consumption of MCT or LCT oil was conducted. During the seven days of daily oil intake, the participants ingested 2x10g oil in 15g cocoa milk on day 1-2, 2x20g oil in 30g cocoa milk on day 3-5, and 2x30g oil in 40g cocoa milk on day 6-7. This corresponded to 812kJ on day 1-2, 1625kJ on day 3-5, and 2413kJ on day 6-7. The participants were instructed to maintain their habitual dietary patterns and physical activity level during the intervention. The participants were instructed to consume the oil together with breakfast and dinner and were supervised to ensure compliance.

After the chronic intake period, a second experimental day (post), mirroring the one of the pre day, was conducted.

After a wash-out period the intervention was repeated in a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 35
* Moderate physical activity level, defined as 1 to 3 weekly sessions of exercise.
* Non-smokers
* No use of medicine
* No known prediabetes or diabetes

Exclusion Criteria:

High habitual intake of MCFA (e.g., coconut milk, coconut oil, or dairy products), A ketogenic diet, known diabetes or pre-diabetes, use of medications, daily use of nicotine products

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Ketone bodies in plasma | Day 0 to day 7
  an increase in plasma ketone bodies induced by intake of medium-chain fatty acids in lean and obese participants

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, D.sci, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark